CLINICAL TRIAL: NCT00265226
Title: Efficacy and Safety Study of Immunomodulator (Mycobacterium w) as an Adjunct Therapy in Category-II Pulmonary Tuberculosis Along With Assessment of Immunological Parameters
Brief Title: Efficacy and Safety Study of Immunomodulator as an Adjunct Therapy in Pulmonary Tuberculosis (TB) Retreatment Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, SK Sharma, Professor and Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-01A/2003-10; NI-705
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2011-07

CONDITIONS: Tuberculosis
Keywords: India; Pulmonary Tuberculosis; Category-II tuberculosis; Immunomodulator; Mycobacterium w; Revised National Tuberculosis Control Programme; Category-II Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — Immuvac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): In one arm the patient will receive intradermal Mycobacterium W Vaccine along with Category II ATT according to RNTCP guidelines
  Interventions: Biological: Intra-dermal administration of Mycobacterium w
- 2 (Placebo Comparator): In this Arm patient will receive Placebo along with Category II ATT drugs according to RNTCP guidelines
  Interventions: Biological: Intra-dermal administration of Mycobacterium w

INTERVENTIONS:
Biological: Intra-dermal administration of Mycobacterium w — Mw Vaccine is given as oral suspension. Total 6 doses are given 0.2 ml at baseline and then 0.1 ml after interval of 2 weeks upto 8 weeks
  Other Names: Immuvac

SUMMARY:
The purpose of the study is to study the efficacy and safety of Mycobacterium in treating patients with lung tuberculosis . Mycobacterium is a strain of bacterium which is used as a vaccine and an adjuvant drug against leprosy. This agent has also been found to be effective in the treatment of lung tuberculosis in a limited number of patients.

The researchers are conducting this study in the World Health Organization (WHO) category-II of lung tuberculosis patients to see the efficacy and also to see any change in immunological parameters.

DETAILED DESCRIPTION:
Mycobacterium w is a recently introduced immunomodulator, which has been found to be useful in rapid killing of Mycobacterium leprae. It improves the clearance of Mycobacterium leprae from the body and is thereby useful in reducing the duration of therapy significantly for multibacillary leprosy. Mycobacterium w shares an antigen with both Mycobacterium leprae as well as Mycobacterium tuberculosis. Mycobacterium w is also found to be useful in the prevention of tuberculosis in experimental animals.

Previous studies on the efficacy of Mycobacterium w as an immunomodulator in pulmonary tuberculosis patients have shown higher sputum conversion rates in patients given Mycobacterium w as an adjuvant therapy along with standard anti-tuberculosis treatment. It has faster and remarkable sputum converting capacity. Similar studies conducted in pulmonary TB category -II [re-treatment as per Revised National Tuberculosis Control Programme (RNTCP), Govt. of India] patients have shown improved cure rates.

Mycobacterium w is commercially available under the brand name of "Immuvac" injection in 0.5 ml multi dose vials approved for use as immunomodulator against Mycobacterium leprae in patients with leprosy. Each vial has 0.5 x 10^9 heat-killed bacilli in a buffered solution. It is manufactured by Cadila Pharmaceuticals Ltd.; Ahmedabad, Gujarat-382 210, India. In this clinical trial one dose consists of 0.1 ml given as an intradermal injection, which contains 10^9 bacilli. A total of 6 doses are given during the Intensive Phase (as per RNTCP, Govt. of India) of treatment. Two injections on both upper arms on day-0 and subsequently one injection on days 14, 28, 42 and 56. No injections are given during the Continuation Phase (as per RNTCP, Govt. of India) of treatment.

As of now, it is not commercially available for use in TB patients as an immunomodulator. Therefore, the investigators are investigating Mycobacterium w (Mw) for its efficacy in TB patients in a "double-blind placebo-controlled randomized clinical control trial" fashion. We are conducting this trial in Category-II pulmonary TB patients (as per RNTCP, Govt. of India), and are assessing the outcome in the form of clinical improvement, sputum conversion and immunological parameters. This is a multi-centric trial sponsored by the Department of Biotechnology, Ministry of Science and Technology, Govt. of India and Cadila Pharmaceuticals Ltd., India.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are sputum positive for pulmonary tuberculosis and who have been treated previously for more than 1 month as per the RNTCP/WHO guidelines.
* Category II inclusion will mean all those patients who are Treatment after Default/Treatment Failure/Treatment Relapse.
* Patients who are willing to give written informed consent.

Exclusion Criteria:

* Patients who are known to be hypersensitive to those ATTs being administered.
* Patients co-infected with HIV, hepatitis B or hepatitis C.
* Pregnant and lactating females or females of child bearing age with a urine HCG positive result 24-48 hours prior to every injection of Mw till 8 weeks.
* Patients with abnormal renal function, liver function or hematological tests.
* Seriously ill and moribund patients with complications such as low lung reserve, marked tachypnoea, chronic cor pulmonale, congestive heart failure.
* Severely malnourished patients with body mass index (BMI) < 15
* Severe hypoalbuminemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1020 (Actual)
Dates: Start 2005-03; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The time of sputum conversion as well as the early sputum conversion between the 2 groups will be evaluated. | from baseline (visit 2)
The cure rate will be evaluated as the primary parameter of efficacy. | 8-9 months
The relapse in patients of category II tuberculosis will be compared in both the groups. | at an interval of 6, 12, 18 and 24 months after the completion of the therapy
Recording of any clinical adverse reactions at anytime during the study for assessment of safety | 2-8 weeks

SECONDARY OUTCOMES:
An additional secondary efficacy endpoint is the patient's and physician's global assessment of the clinical cure. | 8-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, M.D., Ph.D., Study Chair — Professor and Head, Department of Medicine, All India Institute of Medical Sciences, New Delhi, India; Bindu Dey, Ph.D., Study Director — Department of Biotechnology, MST, GOI
Locations (8):
- India (8):
  - Mahavir Hospital, Hyderabad, Andhra Pradesh
  - Smt NHL Municipal Medical College & B.J. Medical College, Ahmedabad, Gujarat
  - National Tuberculosis Institute, Bangalore, Karnataka
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Lala Ram Swarup Institute of Tuberculosis and Respiratory Diseases, New Delhi, National Capital Territory of Delhi
  - SMS Medical College, Jaipur, Rajasthan
  - Tuberculosis Research Centre, Chennai, Tamil Nadu
  - Central JALMA Institute of Leprosy, Agra, Uttar Pradesh

REFERENCES:
- [Background] Patel N, Trapathi SB. Improved cure rates in pulmonary tuberculosis category II (retreatment) with mycobacterium w. J Indian Med Assoc. 2003 Nov;101(11):680, 682. PMID 15198421
- [Background] Patel N, Deshpande MM, Shah M. Effect of an immunomodulator containing Mycobacterium w on sputum conversion in pulmonary tuberculosis. J Indian Med Assoc. 2002 Mar;100(3):191-3. PMID 12408283
- [Background] Katoch K, Katoch VM, Natrajan M, Bhatia AS, Sreevatsa, Gupta UD, Sharma VD, Shivannavar CT, Patil MA, Bharadwaj VP. Treatment of bacilliferous BL/LL cases with combined chemotherapy and immunotherapy. Int J Lepr Other Mycobact Dis. 1995 Jun;63(2):202-12. PMID 7602215
- [Background] Sharma P, Mukherjee R, Talwar GP, Sarathchandra KG, Walia R, Parida SK, Pandey RM, Rani R, Kar H, Mukherjee A, Katoch K, Benara SK, Singh T, Singh P. Immunoprophylactic effects of the anti-leprosy Mw vaccine in household contacts of leprosy patients: clinical field trials with a follow up of 8-10 years. Lepr Rev. 2005 Jun;76(2):127-43. PMID 16038246
- [Background] Sharma P, Kar HK, Misra RS, Mukherjee A, Kaur H, Mukherjee R, Rani R. Reactional states and neuritis in multibacillary leprosy patients following MDT with/without immunotherapy with Mycobacterium w antileprosy vaccine. Lepr Rev. 2000 Jun;71(2):193-205. doi: 10.5935/0305-7518.20000021. PMID 10920614
- [Background] Sharma P, Misra RS, Kar HK, Mukherjee A, Poricha D, Kaur H, Mukherjee R, Rani R. Mycobacterium w vaccine, a useful adjuvant to multidrug therapy in multibacillary leprosy: a report on hospital based immunotherapeutic clinical trials with a follow-up of 1-7 years after treatment. Lepr Rev. 2000 Jun;71(2):179-92. doi: 10.5935/0305-7518.20000020. PMID 10920613
- [Background] Sharma P, Kar HK, Misra RS, Mukherjee A, Kaur H, Mukherjee R, Rani R. Induction of lepromin positivity following immuno-chemotherapy with Mycobacterium w vaccine and multidrug therapy and its impact on bacteriological clearance in multibacillary leprosy: report on a hospital-based clinical trial with the candidate antileprosy vaccine. Int J Lepr Other Mycobact Dis. 1999 Sep;67(3):259-69. PMID 10575405
- [Background] Sharma P, Kar HK, Misra RS, Mukherjee A, Kaur H, Mukherjee R, Rani R. Disabilities in multibacillary leprosy following multidrug therapy with and without immunotherapy with Mycobacterium w antileprosy vaccine. Int J Lepr Other Mycobact Dis. 1999 Sep;67(3):250-8. PMID 10575404
- [Background] Khatri GR, Frieden TR. Controlling tuberculosis in India. N Engl J Med. 2002 Oct 31;347(18):1420-5. doi: 10.1056/NEJMsa020098. PMID 12409545